CLINICAL TRIAL: NCT03302507
Title: Outcomes Following Bilateral Decompression Surgery in Lumbar Spinal Stenosis With Biportal Endoscopy Versus Unilateral Laminotomy Technique: A Prospective, Single-blinded, Randomized Controlled Non-inferiority Trial
Brief Title: Biportal Endoscopy Spine Surgery (BESS )Versus Unilateral Laminotomy Bilateral Decompression (ULBD ): RCT, Non-inferiority Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin S. Yeom, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BESS_001
Record Dates: First submitted 2017-09-21; First posted 2017-10-05 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Degenerative Lumbar Spinal Stenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BESS, biportal endoscopic spine surgery (Experimental): Biportal endoscopic decompression surgery for lumbar spinal stenosis
  Interventions: Procedure: BESS
- ULBD, unilateral laminotomy bilateral decompression (Active Comparator): Minimally invasive ULBD for lumbar spinal stenosis
  Interventions: Procedure: ULBD

INTERVENTIONS:
Procedure: BESS — Biportal endoscopic surgery
  Arms: BESS, biportal endoscopic spine surgery
Procedure: ULBD — Unilateral laminotomy bilateral decompression
  Arms: ULBD, unilateral laminotomy bilateral decompression

SUMMARY:
This study is to compare the clinical outcome between the biportal endoscopic decompression and the unilateral approach bilateral decompression in spinal stenosis

ELIGIBILITY:
Inclusion Criteria:

* patients aged between 30 and 80
* patients who has radiating pain (VAS >=40) on lower extremities with spinal stenosis over Gr B
* patients who required one-level decompression between L1 and S1
* those who (only if a signature was obtainable), or whose legal guardian, fully understood the clinical trial details and signed the informed consent form

Exclusion Criteria:

* Revision surgery
* Over spondylolisthesis Gr II
* Degenerative lumbar scoliosis (Cobb angle >20)
* herniated disc
* patients with a history of other spinal diseases (compression fracture, spondylitis, tumor)
* women with positive pregnancy tests before the trial or who planned to become pregnant within the following 3 years
* patients with a history of malignant tumor or malignant diseases (but the cases of cured disease with no relapse for the past 5 years were included in the present study)
* patients with mental retardation or whose parents or legal guardians were older or had mental disabilities
* other patients viewed as inappropriate by the staff

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Oswestry disability index (ODI) | 3, 6, and 12, months, and every year, up to 5 year after operation
  The ODI is based on a self-administered questionnaire measuring ''back-specific function.'' The questionnaire comprises 10 items, each with 6 levels of response. Each item is scored from 0 to 5, and the total summation is converted to a 0-100 scale. The ODI scores ranges from 0 to 100, with higher scores indicating severe symptoms.
  This is assessed by ODI survey at 1 year after surgery

SECONDARY OUTCOMES:
Visual Analog Pain Scale (VAS) | 4, 8, 12, 24, 48 hours, 2 weeks, 3, 6, and 12, months, and every year, up to 5 year after operation
  VAS is a measurement score that indicates pain severity status. VAS score comprised a 10-cm line with ''none'' (0) on one end of the scale and ''disabling pain'' (10) on the other.
EQ-5D | 3, 6, and 12, months, and every year, up to 5 year after operation
  EQ-5D is a standardized instrument developed by the EuroQol Group as a measure of health-related quality of life that can be used in a wide range of health conditions and treatments. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. This can be used as a quantitative measure of health outcome that reflects the patient's own judgement. The scores on these five dimensions can be presented as a health profile or can be converted to a single summary index number (utility) reflecting preferability compared to other health profiles.
PainDETECT | 3, 6, and 12, months, and every year, up to 5 year after operation
  The painDETECT Questionnaire (PDQ) is a screening tool designed to detect neuropathic pain in patients with chronic low back pain (LBP) based on self-reported pain characteristics. The degree of the seven types of pain quality, the type of pain pattern, and the presence of radiating pain. From the three components of the PDQ, a total score is calculated; a high score indicates that the pain is likely to have a neuropathic component. Scoring is performed using a scoring manual, and results in a final screening score: a score of 0-12 indicates nociceptive pain, 19-38 indicates neuropathic pain, and 13-18 indicates mixed pain.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | up to 1 month after operation
  Surgery related adverse events (incidental durotomy, wound infection, re-operation, re-admission)
Operation duration | Immediate after operation
  Intraoperative time in minutes
Postoperative drainage | Within 3 days after operation
  Total drainage after surgery in milli-liter
Amount of transfusion | Within 7 days after operation
  Total transfusion during and after surgery in milli-liter
Completeness of decompression | Within 3 days after operation
  After surgery, degree of decompression was measured using postoperative MRI
Creatine phosphokinase level in blood | At 2 day after surgery
  Creatine phosphokinase assessment to measure muscle injury at operation
Postoperative Fentanyl consumption | At 3 days after operation
  Total amount of fentanyl consumption after surgery (PCA dose + rescue dose)
Hospital stay | Within 7 days after operation
  Total hospital stay after surgery
Radiographic complications | every year, up to 5 year after operation,
  Disc degeneration, facet degeneration, re-stenosis, back muscle atrophy, kyphotic change, disc rupture
Satisfaction scale | At 1 year after operation
  Satisfaction scale is a short self-report questionnaire for evaluating patient satisfaction with the outcome of lumbar decompression surgery. Items are scored on a 7-point Likert scale with response categories consisting from very satisfied (7 points) to very dissatisfied (1 points).
  Satisfaction after operation at 1 year after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyounggido, South Korea